CLINICAL TRIAL: NCT06757985
Title: Doppler Echocardiography Versus Clinical Targets Guided Therapy on the Outcome of Postpartum Septic Shock, a Randomized Controlled Trial
Brief Title: Doppler Echocardiography Versus Clinical Targets Guided Therapy on the Outcome of Postpartum Septic Shock.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Doppler echocardiography
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Doppler Echocardiography; Postpartum Septic Shock

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTGT group (Experimental): a clinically guided resuscitation protocol, derived from EGDT
  Interventions: Procedure: a clinically guided resuscitation protocol,
- ECHO group (Experimental): a transthoracic bedside focused echocardiographic assessment of the patient
  Interventions: Procedure: a transthoracic bedside focused echocardiographic assessment

INTERVENTIONS:
Procedure: a clinically guided resuscitation protocol, — a clinically guided resuscitation protocol, derived from EGDT and modified to match with the latest survival sepsis campaign guidelines
  Arms: CTGT group
Procedure: a transthoracic bedside focused echocardiographic assessment — a transthoracic bedside focused echocardiographic assessment of the patient will be done, as a baseline ECHO in a three-step approach to monitor hemodynamics using Logiq P7, S5-1 ECHO probe;
  Arms: ECHO group

SUMMARY:
Postpartum sepsis is widely known as a preventable main cause of maternal morbidity and mortality. According to the World Health Organization, approximately 11% of the estimated maternal deaths worldwide were attributed to sepsis. Recent global assessments indicate that obstetric infections rank as the third most prevalent cause of maternal death, with a prevalence mainly observed in low- and middle-income nations.

DETAILED DESCRIPTION:
The management of septic shock is a major medical concern. Early goal-directed therapy emerged as a novel approach for reducing sepsis mortality and was incorporated into Surviving Sepsis Campaign guidelines in 2012. Early detection of sepsis, rapid initiation of antibiotics and effective resuscitation with fluids, vasopressors, and inotropes were important concerns. However, many randomized trials were done to examine the effect of EGDT on morbidity and mortality and showed that EGDT was not associated with a significant reduction in mortality in patients with septic shock compared to usual care. That it wasn't addressed in recent guidelines in 2016 and 2021.

ELIGIBILITY:
Inclusion Criteria:

* postpartum women, within 6 weeks following delivery
* meeting the third international consensus definitions for septic Shock (2016) (Sepsis-3): acute persisting hypotension requiring vasopressors to maintain mean arterial pressure (MAP) ≥ 65 mm Hg and having a serum lactate > 2 mmol/L (18 mg/dL) despite adequate volume resuscitation

Exclusion Criteria:

* Patient refusal
* History of any chronic cardiac disease
* Requirement for immediate surgery
* Hypotension attributable to another cause
* Do-not-resuscitate status
* Contraindication to central venous catheter placement
* Difficult transthoracic echocardiographic evaluation
* Primary cardiogenic cause of shock, instead of sepsis.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
SOFA score | 48 hours.
  The change in Sequential Organ Failure Assessment (SOFA score)

CONTACTS AND LOCATIONS:
Locations (1):
- woman health hospital , Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mouncey PR, Osborn TM, Power GS, Harrison DA, Sadique MZ, Grieve RD, Jahan R, Harvey SE, Bell D, Bion JF, Coats TJ, Singer M, Young JD, Rowan KM; ProMISe Trial Investigators. Trial of early, goal-directed resuscitation for septic shock. N Engl J Med. 2015 Apr 2;372(14):1301-11. doi: 10.1056/NEJMoa1500896. Epub 2015 Mar 17. PMID 25776532
- [Background] Hernandez G, Ospina-Tascon GA, Damiani LP, Estenssoro E, Dubin A, Hurtado J, Friedman G, Castro R, Alegria L, Teboul JL, Cecconi M, Ferri G, Jibaja M, Pairumani R, Fernandez P, Barahona D, Granda-Luna V, Cavalcanti AB, Bakker J; The ANDROMEDA SHOCK Investigators and the Latin America Intensive Care Network (LIVEN); Hernandez G, Ospina-Tascon G, Petri Damiani L, Estenssoro E, Dubin A, Hurtado J, Friedman G, Castro R, Alegria L, Teboul JL, Cecconi M, Cecconi M, Ferri G, Jibaja M, Pairumani R, Fernandez P, Barahona D, Cavalcanti AB, Bakker J, Hernandez G, Alegria L, Ferri G, Rodriguez N, Holger P, Soto N, Pozo M, Bakker J, Cook D, Vincent JL, Rhodes A, Kavanagh BP, Dellinger P, Rietdijk W, Carpio D, Pavez N, Henriquez E, Bravo S, Valenzuela ED, Vera M, Dreyse J, Oviedo V, Cid MA, Larroulet M, Petruska E, Sarabia C, Gallardo D, Sanchez JE, Gonzalez H, Arancibia JM, Munoz A, Ramirez G, Aravena F, Aquevedo A, Zambrano F, Bozinovic M, Valle F, Ramirez M, Rossel V, Munoz P, Ceballos C, Esveile C, Carmona C, Candia E, Mendoza D, Sanchez A, Ponce D, Ponce D, Lastra J, Nahuelpan B, Fasce F, Luengo C, Medel N, Cortes C, Campassi L, Rubatto P, Horna N, Furche M, Pendino JC, Bettini L, Lovesio C, Gonzalez MC, Rodruguez J, Canales H, Caminos F, Galletti C, Minoldo E, Aramburu MJ, Olmos D, Nin N, Tenzi J, Quiroga C, Lacuesta P, Gaudin A, Pais R, Silvestre A, Olivera G, Rieppi G, Berrutti D, Ochoa M, Cobos P, Vintimilla F, Ramirez V, Tobar M, Garcia F, Picoita F, Remache N, Granda V, Paredes F, Barzallo E, Garces P, Guerrero F, Salazar S, Torres G, Tana C, Calahorrano J, Solis F, Torres P, Herrera L, Ornes A, Perez V, Delgado G, Lopez A, Espinosa E, Moreira J, Salcedo B, Villacres I, Suing J, Lopez M, Gomez L, Toctaquiza G, Cadena Zapata M, Orazabal MA, Pardo Espejo R, Jimenez J, Calderon A, Paredes G, Barberan JL, Moya T, Atehortua H, Sabogal R, Ortiz G, Lara A, Sanchez F, Hernan Portilla A, Davila H, Mora JA, Calderon LE, Alvarez I, Escobar E, Bejarano A, Bustamante LA, Aldana JL. Effect of a Resuscitation Strategy Targeting Peripheral Perfusion Status vs Serum Lactate Levels on 28-Day Mortality Among Patients With Septic Shock: The ANDROMEDA-SHOCK Randomized Clinical Trial. JAMA. 2019 Feb 19;321(7):654-664. doi: 10.1001/jama.2019.0071. PMID 30772908